CLINICAL TRIAL: NCT06214689
Title: IDH1 and OCT4 Markers as a Prognostic Factor in Clinical Outcome of High Grade Astrocytic Glioma
Brief Title: IDH1 and OCT4 in High Grade Astrocytoma
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ata Salama Swefy, doctor, Assiut University
Other Study IDs: biomarkers in astrocytoma
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: High Grade Astrocytoma
MeSH Terms: conditions — Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: biomarkers analysis — IDH1 and OCT4 markers analysis of surgical specimens of high grade astrocytoma

SUMMARY:
observation of IDH1 and OCT4 markers level and high grade astrocytoma patients prognosis after excision.

DETAILED DESCRIPTION:
explore the relationship between prognosis and IDH1 and OCT4 biomarkers after high grade astrocytoma excision , according to progression free survival and overall survival , in prospective and retrospective samples.

ELIGIBILITY:
Inclusion Criteria:

* patients of high grade astrocytic glioma patients fit for surgery

Exclusion Criteria:

* patients of low grade glioma patients unfit for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with high grade astrocytic glioma , more than 18 years old and fit for surgery that will be admitted in the department of neurosurgery in Assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
IDH1 and OCT4 markers and their relation to postoperative prognosis of high grade astrocytoma patients | baseline
  explore the relationship between prognosis (progression free and overall survival ) and biomarkers (IDH1 and OCT4 ) after excision of high grade astrocytoma

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine of Assiut University, Asyut, Egypt

REFERENCES:
- [Background] PubMed
- [Result] Ostrom QT, Bauchet L, Davis FG, Deltour I, Fisher JL, Langer CE, Pekmezci M, Schwartzbaum JA, Turner MC, Walsh KM, Wrensch MR, Barnholtz-Sloan JS. The epidemiology of glioma in adults: a "state of the science" review. Neuro Oncol. 2014 Jul;16(7):896-913. doi: 10.1093/neuonc/nou087. PMID 24842956
- [Result] Perry A, Wesseling P. Histologic classification of gliomas. Handb Clin Neurol. 2016;134:71-95. doi: 10.1016/B978-0-12-802997-8.00005-0. PMID 26948349
- [Result] Sathornsumetee S, Rich JN, Reardon DA. Diagnosis and treatment of high-grade astrocytoma. Neurol Clin. 2007 Nov;25(4):1111-39, x. doi: 10.1016/j.ncl.2007.07.004. PMID 17964028